CLINICAL TRIAL: NCT04202016
Title: Three Dimensional Analysis of the Rate of Space Closure With Piezocision-based Corticotomy in Different Facial Types: A Split-mouth Design Randomized Controlled Trial
Brief Title: The Rate of Space Closure With Piezocision-based Corticotomy in Different Facial Types: A Split-mouth Design
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Collaborators: University of Edinburgh (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Hadeel alaathal, Principal Investigator, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 20190232
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Class II Div 1 Malocclusion
Keywords: Canine retraction; Space closure; Rate of tooth movement; Facial divergence; Piezocision
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: The design will be a split-mouth where the participants should need extraction based treatment in collateral sides of the upper arch with one of the sides serving as the treatment while the other will be the control. Then they will be grouped based on their facial type.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A third party will have the randomization of which side to be chosen for each case. An IT student will be asked to prepare randomized two lists using excel Microsoft program. Each list was defined based on facial divergence type; adult high, and adult average lists in the Excel columns. Underneath each list, the raws, equal number of R(right) and L(left) letters will be generated randomly. The orthodontic department's receptionist will receive the excel file, and based on which, prepare closed envelops that will be numbered. Each of which will contain a piece of paper having a letter, either R or L accordingly. The envelops will be dark and difficult to see through even under light. The periodontist will open the envelope of each patient only prior to their piezocision surgery without the involvement of the orthodontist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Piezocision on high facial divergence (Experimental): Piezocision Surgery prior to space closure with closing coil spring four months after extraction. Six weeks later, three other follow up appointments, six weeks apart, taking impressions to measure the rate of space closure.
  Interventions: Procedure: Piezocision Surgery
- High facial divergence (No Intervention): Space closure with coil spring four months after extraction. Six weeks later, three other follow up appointments, six weeks apart, taking impressions to measure the rate of space closure.
- Piezocision on average facial divergence (Experimental): Piezocision Surgery prior to space closure with closing coil spring four months after extraction. Six weeks later, three follow up appointments, six weeks apart, taking impressions to measure the rate of space closure.
  Interventions: Procedure: Piezocision Surgery
- Average facial divergence (No Intervention): Space closure with coil spring four months after extraction. Six weeks later, three other follow up appointments, six weeks apart, taking impressions to measure the rate of space closure.

INTERVENTIONS:
Procedure: Piezocision Surgery — After a surgical cut using #15 surgical blade 2-3 mm distal to the canine a pizocision using piezo-surgery device is made.
  Arms: Piezocision on average facial divergence; Piezocision on high facial divergence

SUMMARY:
23 female participants with class II div I will have extraction of bilateral first bicuspids 10 weeks after bond- up appointment. The extracted teeth will be preserved in special containers for subsequent microscopic analysis. Four months later, upon space closure phase, the patient will have a piezocision surgery on one side randomly chosen. Virtual models will be generated once before the surgery and monthly after for four and a half months. The models will be scanned by CADCAM and later tooth movement will be analyzed in regards to the rugae area.

ELIGIBILITY:
Inclusion Criteria:

* Young adults and adults (15-29).
* Middleastern Caucasian.
* Females.
* Having the defined orthodontic appliance, slot size, prescription, and technique of space closure.
* Class II division I of moderate space requirement that is planned to have the first premolar extracted.
* Average or high facial type.
* Healthy patients without systematic diseases that could affect bone and tooth movement and no contraindication (medical or psychological) to avoid oral surgery.
* No active periodontal diseases as this effect the cytokines expression (stabilized prostaglandin (PG) health)
* Good oral hygiene.
* No other method of non-surgical acceleration technique to be used.

Exclusion Criteria:

* Patients who refused to consent for the study.
* The two extremes of age (younger than 14 and older than 29).
* Having other than the defined orthodontic appliance, slot size, prescription, and technique of space closure.
* Extraction cases of high space requirements or other teeth than the first premolar.
* Patients with systematic diseases that could affect bone and tooth movement and no contraindication (medical or psychological) avoid oral surgery.
* Active periodontal diseases.
* Other methods of non-surgical acceleration technique to be used.

Ages: 15 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of space closure | four and half months
  Every six weeks from the first impression, made on the day of surgery (T0), an impression will be taken, (T1, T2, T3). Images of the impressions will be generated using computer-aided design and computer-aided manufacturing (CADCAM) to evaluate the space changes from a fixed reference point; the rugae area.

SECONDARY OUTCOMES:
Root resorption | Ten weeks
  The extraction will take place 10 weeks after the bonding up-appointment. Atraumatic extraction of the upper first premolars will be executed. The periodontist, performing the extraction, will have the extracted teeth stored in containers that contain sterilized deionized water.
  Each tooth will be placed in ultrasonic bath for 10 minutes to loosen any residual periodontal ligament's and soft tissue fragments' traces which will be later removed by wet gauze with a rubbing motion. Each tooth will be scanned three dimensionally by a desktop X-ray micro-tomography system. Teeth will be scanned with X-rays while being rotated over 360°. Three-dimension object will be generated by a 3D cone beam reconstruction algorithm utilizing the 2D images that have resulted from the scanning process.

CONTACTS AND LOCATIONS:
Overall Officials: Kazem S. Alnimri, Professor, Study Director — Jordan University of Science and Technology
Locations (1):
- Postgraduate orthodontic clinics, Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No